CLINICAL TRIAL: NCT04687579
Title: Elective Umbilical Hernia Repair in Patients With Cirrhosis - a Prospective, Controlled Interventional Study
Brief Title: Elective Umbilical Hernia Repair in Patients With Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Christian Snitkjær, Medical student, Hvidovre University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEROIC21
Record Dates: First submitted 2020-12-21; First posted 2020-12-29 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Cirrhosis, Umbilical Hernia
MeSH Terms: conditions — Fibrosis; Hernia, Umbilical | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical hernia repair (Experimental): Patients with cirrhosis undergoing umbilical hernia repair with or without preoperative optimization. See the section about interventions.
  Interventions: Other: Screening; Procedure: Preoperative optimization; Procedure: Umbilical hernia repair
- Watchful waiting (Other): Patients who do not agree for operation but consent for follow-up. Patients will be followed in the whole inclusion period and can at any time change their preference if they wish to undergo surgery.
  Interventions: Other: Screening

INTERVENTIONS:
Other: Screening — Screening: All health professionals at the hospitals will participate in the screening of umbilical hernia. The screening will be done in the outpatient clinic, the Emergency Department and at the hospital wards.
Procedure: Preoperative optimization — Ascites will be drained using percutaneous drainage or PleurX. Diuretics be used to control ascites preoperative. Haemoglobin < 5 mmol/L indicates the need for red blood cell concentrates using two dosage SAG-M (350-400 mL of red blood cell concentrates in each dose) will be done. Thrombocytopenia < 150 10^9/L will be treated with a TPO-analog using avatrombopag 40-60 mg dispensed as an intravenous fluid. Culture verified infection will be treated with specific antibiotics depending on the blood culture. International Normalized Ratio > 1.7 will be treated with either phytomenadion, Octaplex or fresh frozen plasma depending on the INR.
  Arms: Umbilical hernia repair
Procedure: Umbilical hernia repair — A curved incision placed superiorly or inferiorly around the umbilicus. The umbilicus proper is retained in the skin flap. The blunt dissection is made to the hernia sac. The neck of the herniated sac is then dissected from adjacent tissues by a combination of blunt and sharp dissection. The edges of the fascial defect are measured and the fascial defect is closed with a non-absorbable running suture 2-0. A fitted lightweight polypropylene mesh is placed in an onlay fashion and fixed with 4-8 single non-absorbable sutures in the corners and at the midline, with a mesh overlap of at least 4 cm. The umbilicus is re-inserted with a single knot absorbable suture 3-0. Hemostasis is ensured. Skin closure is performed with Nylon suture 3-0. 20 ml bupivacaine 0.5% is injected to the fascia for early pain control.
  Arms: Umbilical hernia repair

SUMMARY:
Liver cirrhosis is a frequent and severe chronic disease. About 20 % of patients with liver cirrhosis develop umbilical hernias. In comparison, the prevalence in the general population is around 2 %. Patients with liver cirrhosis are often neglected and are not offered equal surgical treatments compared with other patient groups with chronic diseases due to fear of postoperative complications. The current literature is sparse, and many questions remain to be answered, such as timing of repair, risk profile, preoperative staging of the liver disease, possible optimization before surgery, repair technique, and postoperative care. Moreover, nationwide data are lacking.

The management of umbilical hernias in patients with cirrhosis is debated. Recently, European Hernia Society published guidelines stating that elective hernia repair may be safe, and that emergency repair is associated with a high rate of morbidity and mortality. Nonetheless, surgeons remain reluctant to perform elective surgery on these patients due to fear of complications and mortality. The evidence supporting the guidelines is sparse and consists of small, low quality studies. One of the major concerns is that the existing studies failed to use clear and well-described definitions of the underlying severity of the liver disease. The rate of emergency repair may be much higher in patients with liver cirrhosis compared with the general population but there is no data available. The rate of emergency vs elective repair in patients with liver cirrhosis in Denmark is unknown, as well as the rate of reoperation for complications and readmission. Finally, we hypothesize that these patients may benefit from a more proactive approach with early diagnosis of their umbilical hernia by screening, preoperative optimization, and early elective hernia repair, but the effect of this hypothesis needs further evaluation.

ELIGIBILITY:
Inclusion criteria

Patients must meet all the following criteria to be eligible to enrol in the study:

* Age ≥18 years and ≤80 years
* ASA I-III
* Patients with a diagnosis of liver cirrhosis
* Patients with a diagnosis of umbilical hernia (primary or recurrent umbilical hernia)
* Hernia defect size 0,5 cm - 6 cm, only one defect
* Patients who have given written informed consent to participate in the study after having understood this

Exclusion criteria Patients who meet one or more of the following criteria are not eligible to be enrolled in this study

* Patients who cannot cooperate with the trial.
* Patients who cannot read and understand Danish.
* Alcohol- and/or drug abuse - to the discretion of the investigator.
* Fascial gap > 6 cm
* Umbilical hernia repair secondary to another procedure
* If a patient withdraws his/her inclusion consent
* Patients in dialysis

Exclusion from operation

Patients who meet one or more of following criteria on procedure day will not undergo surgery, but can undergo surgery at a later date if none of the criteria are fulfilled:

* ASA IV
* Culture verified infection within two weeks prior to umbilical hernia repair
* Anemia (Hgb < 5?)
* International Normalized Ratio > 1.7
* Thrombocytopenia (<100 mill/mL)
* Large amount of ascitic fluid
* If the operation is considered too risky by any investigator, a patient can always be excluded from surgical intervention based on individual assessment.
* Patients presenting with complicated umbilical hernia (incarceration, rupture, strangulation or ulceration) and the need for acute surgical intervention.
* Patients with BMI > 35 will not undergo surgery. If the patient during inclusion period does not fulfil this criterion (BMI < 35), other exclusion criteria and the rest of inclusion criteria are met then the patient can undergo surgery.
* Thrombolysis within 3 months from umbilical hernia repair

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events | 6 months after umbilical hernia repair and/or inclusion
  1. Death
  2. Life-threatening adverse experience after surgery
  3. Inpatient hospitalization or prolongation of existing hospitalization (for > 24 hours)
  4. Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions

SECONDARY OUTCOMES:
Adverse Events | 6 months after umbilical hernia repair and/or inclusion
  1. A new event which was not pre-existing before intervention.
  2. A pre-existing event which recurs with increased intensity or increased frequency in the follow-up period.
  3. An event which is present at the time of intervention which is exacerbated following initial intervention.

IPD SHARING:
Plan to Share IPD: No